CLINICAL TRIAL: NCT02943733
Title: Safety of TAS-102 in Combination With Temozolomide for Metastatic Pancreatic Neuroendocrine Tumors
Brief Title: Safety of TAS-102 in Combination With Temozolomide for Metastatic Pancreatic NETs
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: closed per sponsor request, for slow enrollment
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16034; NCI-2016-01567 (Registry Identifier: NCI CTRP ID); 2016-0930 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Ver 5.0 12/30/2019 (Other: UW Madison)
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Neuroendocrine Tumors; Neoplasms; Cancer; Tumors
Keywords: Pancreatic neuroendocrine tumors (pNETs); Pancreatic neuroendocrine tumors; pNETs; NETs
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms; Neuroectodermal Tumors, Primitive | interventions — trifluridine tipiracil drug combination; Temozolomide; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS-102 and TMZ (Experimental): Part 1: dose-escalation phase to determine MTD of TAS-102 in combination with Temozolomide (TMZ). Treatment cycles are 28 days, with TAS-102 administered orally twice daily days 1-5 and 8-12, and TMZ administered orally days 8-12. No treatment medications administered days 13-28 of each cycle. Growth factor support is required during Part 1 and should be dosed per institutional standards.
  Part 2: expansion phase to evaluate preliminary efficacy of MTD. Subjects treated with the recommended phase 2 drug doses determined in part 1. Treatment will continue for up to 13 cycles (approx. 12 months). Growth factor support is allowed during Part 2 and should be dosed per institutional standards.
  Interventions: Drug: TAS-102; Drug: Temozolomide; Drug: Filgrastim; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: TAS-102 — Anti-metabolite agent, taken orally.
Drug: Temozolomide — Oral chemotherapy drug.
  Other Names: TMZ
Drug: Filgrastim — Filgrastim provides growth factor support in multiple doses. It stimulates bone marrow to create neutrophils for patients undergoing chemotherapy.
Drug: Pegfilgrastim — Pegfilgrastim provides growth factor support in a single dose. It stimulates bone marrow to create neutrophils for patients undergoing chemotherapy.

SUMMARY:
The goal of this study is to establish maximum tolerated doses/recommended phase 2 dose (RP2D) of temozolomide (TMZ) and TAS-102 when these agents are used in combination and to evaluate the safety profile of this drug combination.

DETAILED DESCRIPTION:
The study is a two part phase 1B clinical trial consisting of three study periods: a screening period of 14 days or less, a treatment period, and a safety follow-up period 30 days after treatment discontinuation.

Part 1 is a dose finding phase with the objective to assess the safety and tolerability of the proposed drug combination and to identify the maximum tolerated dose (MTD) and a recommended phase 2 dose.

Part 2 is an open-label expansion study, which will enroll patients with metastatic pNETs who have not been previously treated with chemotherapy. Part 2 will obtain further safety data of the proposed drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Patients with histologically or cytologically confirmed metastatic or locally advanced NETs of any origin and grade
* Part 1: Presence of evaluable OR measurable disease
* Part 2: Patients with histologically confirmed unresectable or metastatic pNETs of grade 1 or 2.
* Part 2: Presence of measurable disease by RECIST 1.1 criteria
* Concurrent somatostatin analogues are allowed provided that the dose has been stable (+/- 10mg) for at least 8 weeks
* Prior chemoembolization or radiation therapy (including Y90) must be performed at least 2 weeks before study enrollment
* ECOG performance status 0-2
* Life expectancy more than 3 months
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Platelets ≥ 100 x 10^9/L
* AST/ALT ≤ 3 x ULN (≤5 x ULN in case of liver metastases)
* Total serum bilirubin of ≤ x institutional ULN (except for Grade 1 hyperbilirubinemia solely due to a medical diagnosis of Gilbert's syndrome)
* Serum creatinine ≤ 1.5 x institutional ULN (Cockcroft and Gault formula)
* Ability to take oral medication (i.e. no feeding tube)
* Female patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to the start of the study drug treatment and must agree to use adequate birth control if conception is possible during the study and up to 6 months after discontinuation of study drug treatment
* Male patients must agree to use adequate birth control during the study and up to 6 months after discontinuation of study drug treatment
* Women who are nursing must discontinue breast feeding prior to the enrollment in the trial
* Patient must be able and willing to comply with study procedures as per protocol
* Patient able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures

Exclusion Criteria:

* Part 2: Grade 3 tumors or tumors with small cell histology will be excluded
* Previous treatment with TAS-102 or TMZ
* History of partial or total gastrectomy
* Symptomatic CNS metastases requiring treatment
* Prior radiation therapy irradiating more than 10% of total bone marrow
* Other active malignancy requiring treatment within the last 2 years (except for non-melanoma skin cancer, a non-invasive/in situ cancer, or indolent nonmetastatic Gleason 6 prostate cancer)
* Pregnancy or breast feeding
* Active infection requiring treatment
* Known chronic infection with human immunodeficiency virus, hepatitis B, or hepatitis C
* Major surgery within prior 4 weeks (the surgical incision should be fully healed prior to drug administration)
* Any anticancer therapy treatments, including other investigational agents within prior 2 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102 or TMZ
* Extended field radiation within prior 4 weeks or limited field radiation within prior 2 weeks
* Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule
* Ascites, pleural effusion or pericardial fluid requiring drainage in the last 4 weeks
* Uncontrolled diabetes mellitus
* Intestinal obstruction
* Pulmonary fibrosis
* Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure NYHA class III or IV
* Gastrointestinal hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) of TAS-102 | Up to 2 years
  Investigate the safety and determine the MTD of TAS-102 administered in combination with TMZ in patients with advanced NETs. Treatments will continue to disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST).
Part 2: Overall Response Rate | Up to 5 years
  Response rate defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR), assessed as per RECIST criteria. Assessments performed using RECIST criteria.

SECONDARY OUTCOMES:
Part 2: Progression Free Survival (PFS) | Up to 5 years
  Defined as the time from the start of treatment to the date of first documented progression or any cause of death during the study, assessed according to RECIST. Analyzed using the Kaplan-Meier method.
Part 2: Overall Survival | Up to 5 years
  Defined as the time from the start of treatment to the date of expiration. Analyzed using the Kaplan-Meier method.
Part 2: Disease Control Rate | Up to 5 years
  Defined as the percentage of patients who achieved complete response, partial response, and stable disease by investigator assessment as per RECIST.
Part 2: Duration of Response | Up to 5 years
  Analyzed using the Kaplan-Meier method.
Part 2: Safety and Tolerability, Assessed per RECIST Criteria | Up to 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Part 2: Biochemical Response defined as normalization or >50% reduction in levels of Chromogranin A | Up to 5 years
  A major biochemical response will be defined as normalization or >50% reduction in levels of Chromogranin A. Chromogranin A is elevated in up to 60% of functioning and nonfunctioning pancreatic endocrine tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Uboha, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — https://cancer.wisc.edu/